CLINICAL TRIAL: NCT05513963
Title: Feasibility and Effectiveness of the Clairity Tool in a University Mental Health Clinic
Brief Title: Clairity in a University Mental Health Clinic
Acronym: FECU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Clarigent Health (Industry)
Collaborators: Xavier University of Louisiana. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 105-2021
Record Dates: First submitted 2022-03-07; First posted 2022-08-24 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Depression; Anxiety; Suicide; Mental Health Issue
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicide

STUDY DESIGN:
Intervention Model Description: Randomized-Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants will complete a Clairity session between their regular therapy visits. The Clairity interview is between 4-11 minutes where a clinical research coordinator will ask participants questions about hope, secrets, anger, fear, and emotional pain.
  Interventions: Behavioral: Clairity
- Control (No Intervention): Participants will submit demographics and medical records and will only complete standard of care.

INTERVENTIONS:
Behavioral: Clairity — Treatment group participants will complete study session using the Clairity tool in between regularly scheduled therapy visits.
  Other Names: MHSAFE Interview
  Arms: Treatment

SUMMARY:
This is a clinical trial to evaluate the effectiveness of the Clairity tool within the university setting for students who are being seen by a mental health provider.

DETAILED DESCRIPTION:
In this study, the investigators plan to evaluate the effect of the Clairity process in a university setting. The Clairity process will be implemented as a 15-20 minute "between-the-visit" mental health check-in between a patient and clinical staff. Clairity will record and analyze patient speech using artificial intelligence algorithms developed for early detection and monitoring of mental health and suicidal risk. This study will be the first to return Clairity results real time to the clinician. The study employs a mixed-methods design, using rolling recruitment of clients of the Xavier University Psychological services clinic (XUPS) during the 2022-2023 school year. Study-trained clinical research coordinators will begin enrolling participants after completing the online protocol training and brief human subject's protection training.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Currently a client receiving services from XUPS
* Able to provide informed consent
* Speaks and understands English fluently
* Willing to abide by all research procedures

Exclusion Criteria:

* Participants with communication disorders (linguistic or articulation) or who cannot articulate clearly in English.
* Participants with an intellectual and/or neurocognitive disability that the study staff deems a barrier to participation.
* History of any other serious medical or psychiatric condition that would interfere with the ability of the patient to complete the study or would make it ethically unfeasible to enroll.
* Any participant, who at the discretion of the study staff, should not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11-03 (Estimated)

PRIMARY OUTCOMES:
Clairity Dashboard | 12 month
  A clinical dashboard (Clairity) where consolidated results of standardized instruments and language-based machine learning models can more fully inform and expedite the clinical decision-making process. This type of dashboard can provide the clinician a time-based snapshot of the current mental state of the client and can inform the clinician of whether treatment methods are making an impact. The addition of an unbiased, innovative measure derived from vocal biomarkers may bring objectivity to the current methods. Multiple data points for a client's session displayed in the Clairity dashboard will support the clinician's ability to reliably monitor clients' progress and make more informed and reliable clinical decisions.
Identify Mental States with Area Under the AUC metric | 12 month
  The area under the receiver operating characteristic (AUC) metric is popular when evaluating machine learning models because it does not impose arbitrary thresholds for classification, as is required for other metrics, such as sensitivity and specificity. An AUC of 0.5 is a model that predicts as well as random chance, and an AUC of 1.0 is a perfect model. In the social sciences, an AUC ≥ 0.8 is considered excellent. An AUC ≥ 0.8 for suicidal risk and depression will be the target. To meet this target with tolerances for type I (α) and type II (β) errors at 0.01 and 0.95 respectively, and an allocation ratio of 1 (number of controls/number of cases), a sample size analysis determines 25 cases and 25 controls for each condition. While many of the conditions of interest exist as comorbidities, historical data at the XUPS clinic supports a sample of 50 clients measured over four interactions will meet the required case-control numbers for each condition.
Outcome Measure Comparison | 12 month
  To measure the potential impact of the Clairity process, clients will complete their treatment as usual, which includes the Outcome Questionnaire-45 (OQ-45) prior to therapy sessions. The OQ-45 is a quantitative self-report inventory used to assess therapy progress. A repeated measures ANOVA will be used to compare scores on the OQ-45 for control and treatment participants enrolled in the study over an eight-week treatment period. Additionally, changes to treatment plans and therapy attendance between the two groups will be examined.
Clinical Utility Treatment Outcomes | 12 month
  Additional mental health data collected through Clairity, delivered via a dashboard, will provide value to clinicians that may influence therapy, such as altering treatment plans or creating safety plans. Qualitative survey data will be collected to understand how clinicians use and value this information. An evaluation of the change in clients' scores over time on the Outcome Questionnaire-45 for those in the control and treatment groups will also occur. This will allow the investigators to estimate the effect, if any, the Clairity process has on clients' mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- Xavier University Psychological Services Clinic, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided